CLINICAL TRIAL: NCT04678713
Title: Maximal Fat Oxidation and Fuel Use During Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Deakin University (Other)
Responsible Party: Principal Investigator, Jørn Wulff Helge, Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Variation in MFO
Record Dates: First submitted 2020-11-13; First posted 2020-12-22 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Obesity
Keywords: Maximal fat oxidation; Ketogenic diet; Carbohydrate rich diet; Fat rich diet; Maximal aerobic capacity; Trained individuals; Adipose triglyceride lipase; The maximal fat oxidation intensity; Glucose Transporter 4; Citrate synthase; Hydroxyacyl-Coenzyme A dehydrogenase; Hormone sensitive lipase; Intramuscular Triacylglycerol; Respiratory exchanges ratio; Glycogen synthase; Hexokinase II
MeSH Terms: conditions — Obesity; Wolman Disease

STUDY DESIGN:
Intervention Model Description: The participants will be separated into 2 groups by stratified randomization consuming either a Fat rich diet (HiFAT) or a carbohydrate rich diet (HiCHO) (n=40 in total).
  When all 40 participants have completed the study, the results will be analysed by separating the two groups into two subgroups based on the median of the MFO
Masking Description: As the participants receive a specific diet, and have to buy their gloceries themself, it is not possible to mask what kind of diet they consume. They will be randomised into what kind of diet they receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fat rich diet (Experimental): Participants consuming 3 days of fat rich diet
  Interventions: Dietary Supplement: investigate the nutritional determinants of MFO in moderate to well-train individuals; Other: Investigate the physiological determinants of MFO in moderate to well-train individuals
- Carbohydrate rich diet (Experimental): Participants consuming 3 days of carbohydrate rich diet
  Interventions: Dietary Supplement: investigate the nutritional determinants of MFO in moderate to well-train individuals; Other: Investigate the physiological determinants of MFO in moderate to well-train individuals

INTERVENTIONS:
Dietary Supplement: investigate the nutritional determinants of MFO in moderate to well-train individuals — The participants will receive a 3-day fat rich or a carbohydrate rich diet. The participants will perform a maximal fat oxidation test before and after the diet intervention to evaluate the effect of the two diets on MFO.
Other: Investigate the physiological determinants of MFO in moderate to well-train individuals — Muscle biopsies will be obtained at baseline to compare muscle characteristics between well-matched train individuals with a high compared to a low maximal fat oxidation.

SUMMARY:
Fat and carbohydrate are the two main energy stores available as fuel during exercise. It is well known that the exercise intensity and feeding status are the major factors determining the type of fuel used during exercise. During prolonged exercise at low to moderate exercise fat is the primary fuel being used and to improve performance studies has tried to understand strategies to maximize muscle glycogen storage and elevate fat oxidation during exercise. With this strategy they aim for preserving the limited muscle glycogen stores and thus improving endurance performance. In relation to this the maximal fat oxidation (MFO: The highest rate of fat oxidation across all exercise intensities) has been studied as increasing the fat oxidation could decrease the depletion of the glycogen stores. Further it has recently been shown that MFO is related to performance in endurance trained. However the MFO has been found to vary markedly between trained individuals matched on their activity level.

It has been suggested that the diet and subsequent substrate availability during exercise contributes independently to the variation in MFO. However, the measurements have never been evaluated in a trained group with similar aerobic capacity and training status. Therefore, the aim of the study is to investigate the effect of a short term fat rich or carbohydrate rich diet on MFO in well trained men with a high vs. a low MFO. The hypothesis is that 3 days of a fat-rich diet will increase MFO while 3 days of a Carbohydrate rich diet will decrease MFO in both individuals with a high MFO (HiMFO) and a low MFO (LoMFO). Furthermore, it is hypothesized that HiMFO will have a significantly higher MFO after both diets compared to LoMFO.

Lifestyle and physiological factors have been investigated to determine the variation of the MFO capacity. However, these factors can only explain 50% of the interindividual variability in MFO. Despite the critical role of fat oxidation during exercise, few studies have explored the differences in skeletal muscle characteristics between HiMFO and LoMFO. The second aim of the study is thereby to investigate if muscle characteristics can explain the variability in MFO within well-trained males. The hypothesis is that HiMFO will have more favorable muscle characteristics for fat oxidation compared to LoMFO including a higher oxidative capacity, intramuscular triacylglycerol concentration and a higher expression of key enzymes in lipid metabolism.

DETAILED DESCRIPTION:
A group of young, healthy and moderate to well-trained males will be recruited for the study. The participants will be separated into 2 groups by stratified randomization consuming either a 3 day Fat rich diet (HiFAT) or a carbohydrate rich diet (HiCHO).

When all participants have completed the study, the results will be analysed by separating the two groups into two subgroups based on the median of the MFO

The study includes 4 visits to out laboratory.

When the participants have read, accepted and signed the plain language statement they will be invited for a screening session in our laboratory which is the first visit. If the participant meet the inclusion and not the exclusion criteria, they will be included in the study and a time schedule for the next three visits will be planned. In the end of the screening the participant will be instructed to full fill a 4-day diet dairy to analyse the participants habitual diet.

For the second visit the participant will meet in the laboratory after an overnight fast and has been asked to avoid alcohol and strenuous exercise 48 hours prior to the test day. The second test starts with a visit to the toilet before a Dual-energy X-ray absorptiometry (DXA) scan and a bioelectrical impedance scan (BIA) is performed to measure the body composition of the participant. After 5 min. of rest, the blood pressure is measured followed by a measurement of the hip and waist circumference. After measuring the blood pressure and body composition the participant will perform a incremental exercise test on a cycle ergometer. The expired air is measured by indirect calorimetry and is used to calculate the maximal fat oxidation and maximal aerobic capacity.

As the second visit, the participant will arrive to laboratory in the morning after an overnight fast having been asked to avoid alcohol and strenuous exercise 48 hours prior to the test day. At the third visit a resting blood samples, fat and muscle biopsies are collected. After 30 min. of rest the same incremental exercise test will be performed as at visit 2 to measure the maximal fat oxidation and maximal aerobic capacity. The test is performed twice to minimize the variation and to ensure the circumstances with the biopsies are identical before and after the diet intervention.

At the end of the third visit, the participant will receive a high fat or isoenergetic high carbohydrate diet to follow for the next three days. The participant will further receive an activity watch to track his activity level during the diet intervention and he will be instructed to exercise for one hour at 65 % of his maximal heart rate.

The fourth and last visit to the laboratory is the day after finishing the three days diet intervention. The participant arrive to laboratory in the morning after an overnight fast having been asked to avoid alcohol and strenuous exercise 48 hours prior to the test day. The test day initiates with a visit to the toilet to empty the bladder and a DXA and BIA are performed followed by a measurement of the blood pressure and the hip and waist circumference. The participant is led to the laboratory where he has to rest for 5-10 min. before collecting a resting blood sample and a fat and muscle biopsy. The participant has to rest for further 30 min. before performing the incremental exercise test to measure the maximal fat oxidation and maximal aerobic capacity.

Procedure and analysis:

Blood samples: The blood samples will be collected from the vein cubiti medialis in the forearm. The blood samples will be analyzed using a standard lab biochemical assays to assess metabolic risk factors and plasma metabolites and hormones.

Fat biopsy: The fat biopsies will be collected from the abdominal subcutane adipose tissue 3-5 cm. lateral from the navel. The samples will be collected by the Bergstrom biopsy technique using a Bergstrom biopsy needle. The fat biopsy will be analysed using microscopy and High Resolution Mitochondria Respirometry to assess the mitochondria capacity, the inflammation of the macrophage and the size of the adipose cells. Furthermore, the expression of proteins and enzymes important for the glucose and fat metabolism will be measured.

Muscle biopsy: The muscle biopsies will be collected from musculus vastus lateralis by the doctor of our department using the Bergstrom biopsy technique. The muscle biopsy will be analysed by immunofluorescence microscopy and the Western blot technique to assess muscle characteristics (e.g muscle fibre type, capillary density and fibre type specific IMTG content) and the expression of key proteins involved in FFA uptake, intramuscular lipolysis and fat oxidation.

The expected outcomes This study will help us to understand the underlying muscular mechanism explaining why substrate use is different amongst a group of similar well-trained athletes. The study will further illuminate if individuals with a high maximal fat oxidation react differently to a high fat or carbohydrate diet compared to individuals with a low maximal fat oxidation.

This information will be highly relevant for coaches, federations, nutritionists and endurance trained athletes looking to optimize nutritional and training methods to enhance metabolic responses and ultimately improve exercise performance.

Statistical analysis:

A Pearsons correlation analyse was performed including all relevant physiological variables regarding the primary outcome, Maximal fat oxidation to analyse the physiological differences between the group with a high MFO and low MFO.

Furthermore a two way ANOVA with repeated measurements will be performed to analyse any effect of the diet on MFO and to analyse if there is any differences on the effect of diet between individuals with a high compared to low MFO. Any significant effects from the ANOVA test will be analysed with a post hoc test to evaluate the interaction between HiMFO and LoMFO.

The significant level is p<0.05.

General design:

The project was approved by the Science Ethical commitee of the greater region of Copenhagen (H-20019103) the 3rd of July 2020. The protocol of the study adhered to the principles of the Helsinki declaration.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 40 years
* Physical activity > 3 times/week
* Maximal aerobic capacity > 50 mlO2/min/kg
* BMI < 30 kg/m2

Exclusion Criteria:

* Aged below 18 years or above 40 years
* Maximal aerobic capacity < 50 mlO2/kg/min
* Body mass index > 30 kg/m2
* Taking any prescription medication influencing metabolism
* Having existing cardiovascular, metabolic or musculoskeletal conditions that may influence ability to exercise or study outcomes

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Change in maximal fat oxidation | Baseline and after three days diet
  Change in maximal fat oxidation (gram/min.) from baseline to after 3-day carbohydrate rich or fat rich diet in moderately trained males

SECONDARY OUTCOMES:
Change in muscle triacylglycerol | Baseline and after three days diet
  Change in muscle triacylglycerol (arbitrary unit) from baseline to after 3-day carbohydrate rich vs. fat rich diet in moderately trained males

CONTACTS AND LOCATIONS:
Overall Officials: Jørn Helge, Professor, Principal Investigator — Department of Biomedical Sciences, Faculty of Health and Medical Sciences, University of Copenhagen
Locations (1):
- Xlab, Faculty of Health and Medical Sciences, University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No